CLINICAL TRIAL: NCT06798974
Title: Effect of Three-Dimensional Lemon Video on Thirst Perception and Dehydration-Related Discomfort in Intensive Care Unit Patients Undergoing Colorectal Surgery: Randomized Controlled Study
Brief Title: Effect of Three-Dimensional Lemon Video on Thirst Perception and Dehydration-Related Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Serpil SU, Lecturer, PhD, RN, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NecErUniveristy
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Thirst in Intensive Care Unit (ICU) Practice

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three-dimensional video (Experimental)
- Control (No Intervention)

INTERVENTIONS:
Other: Three-dimensional video — Patients who meet the criteria for inclusion in the study will be randomly assigned to intervention and control groups. The intervention group will be shown a 3D lemon video with virtual reality glasses. The video will be created by a company that shoots 3D videos. Opinions of three experts will be obtained for the suitability of the video. The video will be shown to patients for 5 minutes. In order to control the effects that may arise from the practitioner during the study, the virtual reality glasses application will be applied to all patients by the same clinic nurse. The control group will not receive any intervention and will receive standard care. Data collection forms will be given to the patient by the researcher and will be collected after the patient fills them out.

SUMMARY:
This study will be conducted to investigate the effects of a three-dimensional lemon video shown to intensive care patients undergoing colorectal surgery on thirst perception and thirst-related discomfort. The study will be conducted as a randomized controlled, single-blind experimental design. The universe of this study, which will be conducted in the General Surgery Intensive Care Unit of the Necmettin Erbakan University Medical Faculty Hospital, will consist of volunteer patients who will be admitted to the intensive care unit. The sample of the study will consist of 70 patients. In the study, patients will be divided into two groups as virtual reality glasses and control groups. The virtual reality glasses group will be shown a three-dimensional lemon video. Standard care will be provided to patients in the control group. Patients will be assigned to the groups using the block randomization method. Randomization will be performed using a random number table in a computer environment (www.random.org). Research data will be collected using the Descriptive Characteristics Form, Numerical Rating Scale, and Surgical Period Thirst-Related Discomfort Scale (CDSBRÖ). Ethics committee approval and institutional permission will be obtained before collecting research data. Appropriate statistical tests will be used in the evaluation of the data.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65,
* Those who have undergone colorectal surgery,
* Those who are oriented to time and place,
* Those who are literate,
* Those who have been admitted to the general surgery intensive care unit,
* Those who are being monitored in the postoperative period,
* Those who volunteer to participate in the study,
* Those who can communicate verbally,
* Those who are open to communication and cooperation,
* Those who do not have visual and auditory impairments,
* Those who do not use glasses or have no visual impairments,
* Those who do not have cognitive-psychological disorders,
* Those who are not diagnosed with renal failure,
* Those who do not have oral intake according to the physician's order,
* Those who are not connected to a mechanical ventilator will be included in the study.

Exclusion Criteria:

* Patients who have undergone a second surgical procedure during their hospitalization,
* Patients who have open wounds on their mouth or lips,
* Patients who have been diagnosed with migraine or vertigo,
* Patients who have nausea and vomiting will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale | The 1st measurement will be made immediately before watching the 3D video, the 2nd measurement will be made within 1 minute after watching the 3D video, and the 3rd measurement will be made 30 minutes after watching the 3D video.
  It will be used to assess the intensity of thirst perception. This scale has numerical values between 0-10 points and the individual is shown the scale and asked to choose the number that best describes thirst. It consists of a horizontal line that starts with the expression "0" or "I'm not thirsty at all" and ends with the expression "10" or "I'm very thirsty".
Perioperative Thirst Discomfort Scale | The 1st measurement will be made immediately before watching the 3D video, the 2nd measurement will be made within 1 minute after watching the 3D video, and the 3rd measurement will be made 30 minutes after watching the 3D video.
  The scale is a 3-point Likert-type scale consisting of 7 items including dry mouth, dry lips, swollen tongue, saliva density, dry throat, bad taste in the mouth and desire to drink water. Rating is done as; It did not bother (0), It bothered a little (1) and It bothered a lot (2). The scale has no sub-dimensions. The lowest score from the original scale total is 0 and the highest is 14. The expression "Skewered slice" from the scale items was removed from the Turkish scale because it had a low factor load. The lowest score from the scale total is 0 and the highest is 12. Higher scores indicate more thirst.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No